CLINICAL TRIAL: NCT01094743
Title: Dispensing Evaluation of a Prototype Contact Lens and a Marketed Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-1636AZ
Record Dates: First submitted 2010-03-24; First posted 2010-03-29 (Estimated); Results first posted 2012-01-25 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- galyfilcon A prototype lens / lotrafilcon B lens (Other): The galyfilcon A prototype lenses will be worn during the first period and lotrafilcon B lenses will be worn during the second period. Each period consists of daily lens wear for one week.
  Interventions: Device: galyfilcon A prototype lens; Device: lotrafilcon B lens
- lotrafilcon B lens / galyfilcon A prototype lens (Other): The lotrafilcon B lenses will be worn during the first period and galyfilcon A prototype lenses will be worn during the second period. Each period consists of daily lens wear for one week.
  Interventions: Device: galyfilcon A prototype lens; Device: lotrafilcon B lens

INTERVENTIONS:
Device: galyfilcon A prototype lens — Silicone hydrogel contact lens
Device: lotrafilcon B lens — Silicon Hydrogel contact lens

SUMMARY:
The purpose of this study is to compare visual acuity and redness of eyes between a prototype contact lens and an already marketed contact lens.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be at least 18 years of age and no more than 39 years of age.
2. The subject is a current spherical soft contact lens wearer (defined as a minimum of 6 hours of DW for a minimum of 1 month prior to the study) and willing to wear the study lenses on a daily wear basis (defined as a minimum of 6 hours of wear per day at least five days of the week) for the duration of the study.
3. The subject's optimal vertexed spherical equivalent distance correction must be between -1.00 and - 9.00D.
4. Any cylinder power must be ≤ -0.75D.
5. The subject must have visual acuity best correctable to 20/25+3 or better for each eye.
6. The subject must read and sign the Statement of Informed Consent.
7. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.

Exclusion Criteria:

1. Ocular or systemic allergies or disease which might interfere with contact lens wear.
2. Systemic disease or use of medication which might interfere with contact lens wear.
3. Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.
4. Clinically significant (grade 3 or 4) tarsal abnormalities or bulbar injection which might interfere with contact lens wear.
5. Any ocular infection.
6. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
7. Pregnancy or lactation.
8. Diabetes.
9. Infectious diseases (e.g. hepatitis, tuberculosis) or an immuno-suppressive disease (e.g. HIV).
10. Habitual contact lens type is toric, multifocal, or is worn as extended wear.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2010-03-01 (Actual); Study Completion 2010-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Jacksonville, Florida
  - Salem, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Galyfilcon A Prototype Lens / Lotrafilcon B Lens: All enrolled subjects were to wear both lenses through the course of the study.
Period: Period 1
Arm/Group | Galyfilcon A Prototype Lens / Lotrafilcon B Lens
Started | 52
Completed | 50
Not Completed | 2
Not completed — Unsatisfactory comfort at lens fitting | 2
Period: Period 2
Arm/Group | Galyfilcon A Prototype Lens / Lotrafilcon B Lens
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Galyfilcon A Prototype Lens / Lotrafilcon B Lens
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (5.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 35
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity Monocular
Description: Snellen monocular visual acuity measurement
Time Frame: after 1 week of lens wear
Population: All completed subjects
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Groups:
- Galyfilcon A Prototype: All subjects who wore the galyfilcon A prototype lens; VA measured after one week of daily contact lens wear.
- Lotrafilcon B: All subjects who wore the lotrafilcon B lens; VA measured after one week of daily contact lens wear.
Arm/Group | Galyfilcon A Prototype | Lotrafilcon B
Number analyzed (Participants) | 50 | 50
Number analyzed (eyes) | 100 | 100
eyes
  20/15 monocular | 59 | 64
  20/20 monocular | 40 | 30
  20/25 monocular | 1 | 5
  20/30 monocular | 0 | 1

2. Primary Outcome: Visual Acuity Binocular
Description: Snellen binocular visual acuity measurement
Time Frame: after 1 week of lens wear
Population: All completed subjects
Measure: Number; unit: participants
Arm/Group | Galyfilcon A Prototype | Lotrafilcon B
Number analyzed (Participants) | 50 | 50
participants
  20/15 binocular | 40 | 42
  20/20 binocular | 10 | 8

3. Primary Outcome: Subjective Assessment of Lens Comfort
Description: Contact Lens User Experience (CLUE)TM questionnaire: A validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response.
Time Frame: after 1 week of lens wear
Population: Completed subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galyfilcon A Prototype | Lotrafilcon B
Number analyzed (Participants) | 50 | 50
units on a scale | 66.23 (24.112) | 55 (21.844)

4. Secondary Outcome: Limbal Redness
Description: Scale of 0 to 4, where 0=None, 2=Trace, 3=Mild, 4=Moderate, 5=Severe.
Time Frame: after 1 week of lens wear
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Galyfilcon A Prototype | Lotrafilcon B
Number analyzed (Participants) | 50 | 50
Number analyzed (eyes) | 100 | 100
eyes
  Grade 0 None | 37 | 35
  Grade 1 Trace | 61 | 61
  Grade 2 Mild | 2 | 4

5. Secondary Outcome: Bulbar Redness
Description: Scale of 0 to 4, where 0=None, 2=Trace, 3=Mild, 4=Moderate, 5=Severe.
Time Frame: after 1 week of lens wear
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Galyfilcon A Prototype | Lotrafilcon B
Number analyzed (Participants) | 50 | 50
Number analyzed (eyes) | 100 | 100
eyes
  Grade 0 None | 44 | 34
  Grade 1 Trace | 50 | 64
  Grade 2 Mild | 6 | 2

6. Primary Outcome: Subjective Assessment of Quality of Vision
Description: as for outcome 3
Time Frame: after 1 week of lens wear
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galyfilcon A Prototype | Lotrafilcon B
Number analyzed (Participants) | 50 | 50
units on a scale | 63.22 (25.345) | 59.83 (20.036)

7. Secondary Outcome: Subjective Assessment of Lens Comfort
Description: as for outcome 3
Time Frame: 10 minutes after lens insertion at time of initial lens fitting
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galyfilcon A Prototype | Lotrafilcon B
Number analyzed (Participants) | 50 | 50
units on a scale | 76.67 (18.487) | 65 (19.842)

ADVERSE EVENTS:
Arm/Group | Galyfilcon A Prototype Lens / Lotrafilcon B Lens
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication requires agreement and written consent from the Sponsor.